CLINICAL TRIAL: NCT07376187
Title: Digital Physiotherapy Services in the Management of Pediatric Chronic Suppurative Lung Diseases: A Randomized Controlled Trial
Brief Title: Digital Physiotherapy for Pediatric Chronic Suppurative Lung Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Aspasia Mavronasou, PT, MSc, PhD candidate, Principal Investigator, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22510/25
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Suppurative Lung Disease; Protracted Bacterial Bronchitis; Primary Ciliary Dyskinesia (PCD); Non Cystic Fibrosis Bronchiectasis
Keywords: chronic suppurative lung diseases; digital health services; pediatric; physiotherapy; remote; website
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Intervention Model Description: Two-arm (1:1), single blinded, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Block Randomisation, Initial and final outcome assessors blinded to treatment arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Health Services Group (DHSG) (Active Comparator): The treatment arm will receive a home-based hybrid (synchronous and asynchronous) remotely administered exercise program and ACTs for 12 weeks. Children will perform ACTs daily and will participate in an exercise program. The exercise program will consist of 16 exercises per session, varied on the four-letter words chosen at a time. At each session, a combination of four words will be performed and modified weekly. Additionally, they will have access to a website for disease management, including information about common symptoms, nutrition, pharmacological treatment, exercise, and ACTs performance. They will receive via website automated weekly reminders for ACTs and exercise performance, and can report daily symptomatology and track any clinical fluctuations.
  Interventions: Device: Videoconferencing (Vsee platform); Device: Specially designed website (FysΑΩ)
- Control Group (CG) (No Intervention): Participants in the control group will receive usual care, typically comprising inhaled antibiotics and/or bronchodilators for respiratory infections as regular pharmacological treatment in clinically stable condition and a 40-minute, in-person, physiotherapy session where they will be taught ACTs to perform at home. A printed copy of a handbook, including information on their disease and symptoms, nutrition, pharmacological treatment, exercise, and how to perform airway clearance techniques, will be provided.

INTERVENTIONS:
Device: Videoconferencing (Vsee platform) — The prescribed weekly regimen will consist of 50-minute remote sessions: two synchronous, supervised sessions conducted via the Vsee platform, and a minimum of one asynchronous, unsupervised session. Children will perform ACTs (including individualized teaching and review of postural drainage, percussion, vibration, ACTs devices, huffing, coughing), diaphragmatic breathing, and blowing games. During the synchronous, supervised videoconference sessions, they will be monitored/supervised by the pediatric physiotherapist. The exercise program will be based on the 24-letter Greek alphabet, where each letter represents an individual aerobic or strengthening exercise. The exercise program consists of 16 exercises per session, varied on the four-letter words chosen at a time. At each session, a combination of four words will be performed. The exercise program will last 25 to 30 minutes per session. The exercise workload will be equal to 60 - 70% of maximum heart rate.
  Arms: Digital Health Services Group (DHSG)
Device: Specially designed website (FysΑΩ) — The DHSG will be granted access to a website (www.fysao.gr) for disease management, including information about common symptoms, nutrition, pharmacological treatment, exercise, and ACTs performance. To facilitate adherence and longitudinal monitoring, the DHSG will receive automated weekly reminders for ACTs and exercise performance. Through the web portal's integrated evaluation forms, children can report daily symptomatology and track any clinical fluctuations. All the ACTs and the exercise program have been digitized as high-definition videos and images, ensuring asynchronous accessibility for the DHSG. Furthermore, the platform facilitates secure communication, enabling children and their parents/caregivers to communicate with healthcare professionals via integrated email or direct document transmission.
  Arms: Digital Health Services Group (DHSG)

SUMMARY:
This is a prospective, single-center, two-arm (1:1), assessor-blinded, randomized controlled clinical trial that will be conducted in collaboration with the outpatient clinic of the third Pediatric Pulmonology Unit, "Attikon" University Hospital of Athens in Greece. The aim of the study is to investigate the effects of applying digital physiotherapy services in the management of specific clinical outcomes in children with chronic suppurative lung diseases, other than cystic fibrosis. The research question is whether airway clearance techniques and exercise training that are performed remotely using digital health services (DHSs) can improve functional and exercise capacity, as well as compliance with ACTs, compared to usual care. The intervention program includes airway clearance techniques (ACTs), as well as aerobic and strengthening exercises that can be implemented easily in an online setting at home with minimal equipment. The duration of the program will be 12 weeks, and the prescribed weekly regimen will consist of 50-minute remote sessions: two synchronous, supervised sessions conducted via the Vsee platform, and a minimum of one asynchronous, unsupervised session. Children will be encouraged to maintain daily adherence to the exercise protocol.

DETAILED DESCRIPTION:
This is a prospective, single-center, two-arm (1:1), assessor-blinded, randomized controlled clinical trial that will be conducted in collaboration with the outpatient clinic of the third Pediatric Pulmonology Unit, "Attikon" University Hospital of Athens in Greece. The aim of the study is to investigate the effects of applying digital physiotherapy services in the management of specific clinical outcomes in children with chronic suppurative lung diseases, other than cystic fibrosis. The collection of medical history will be conducted via a 40-minute synchronous videoconference session. Children will be randomized into parallel arms: the digital health services group (DHSG) and the control group (CG). All children will receive usual care, including inhaled antibiotics and/or bronchodilators for respiratory infections, alongside recommendations to maintain regular physical activity and to perform ACTs. Furthermore, all child-parent/caregiver dyads will attend a 40-minute, in-person session with the physiotherapist at the outpatient clinic. This session is designed to provide standardized training on airway clearance techniques (ACTs) for subsequent implementation at home. The DHSG will undergo a 12-week home-based hybrid (synchronous and asynchronous), remotely administered exercise program and ACTs. Likewise, the DHSG will have access to a specifically designed website about disease management (www.fysao.gr). The intervention program includes airway clearance techniques (ACTs), as well as aerobic and strengthening exercises that can be implemented easily in an online setting at home with minimal equipment. The prescribed weekly regimen will consist of 50-minute remote sessions: two synchronous, 1:1 supervised sessions conducted via videoconferencing, and a minimum of one asynchronous, unsupervised session. All outcome measures will be assessed at the following time points: baseline (before the intervention), the end of the intervention (12 weeks), and follow-up (6 months after the intervention has ended). All clinical assessments will be conducted in-person at the outpatient clinic by blinded healthcare professionals. Changes from baseline in functional and exercise capacity, compliance with ACTs, respiratory and peripheral muscle strength, physical activity and sedentary behavior, as well as quality of life, will be assessed at 3 and 6 months for both groups.

ELIGIBILITY:
Inclusion Criteria

* children aged 6 to 12 years old
* clinically stable with an absence of pulmonary exacerbation four weeks prior to the study's recruitment
* adherence to attend regular medical follow-up from a pediatric pulmonologist every three months

Exclusion Criteria:

* Cystic fibrosis
* Immunodeficiency or asthma as their primary condition
* Clinical evidence of cardiovascular, neuromuscular, metastatic, or psychiatric comorbidities, and neuromuscular or musculoskeletal impairments that affect mobility and the ability to follow instructions
* Medical history of lung transplant
* Participation in other rehabilitation programs, or attendance at regular physiotherapy ACTs sessions (>10 sessions in a 3-month period)
* Lack access to the internet (e.g., no smartphone, tablet, or laptop)
* Inability to use technological devices

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity (modified Shuttle Walk test) | Change From Baseline in MSWT distance at 3 and 6 months
  Maximal exercise capacity will be assessed through the modified shuttle walk test (MSWT). In the MSWT, participants will be asked to walk rapidly at gradually increasing speeds (15 levels total) along a 10-m corridor. An audio signal ("beep") will mark the transitions between levels, signaling a required increase in velocity. The protocol will commence at a baseline speed of 0.5 m/s (Level 1), with an incremental increase of 0.17 m/s for each subsequent level. The test will be terminated based on inability to continue, symptomatic fatigue, or the failure to reach the course marker before the auditory signal on two consecutive occasions. The walking distance (MSWD) will be recorded. Two trials will be performed, with at least a 30-minute rest.
Compliance with the airway clearance techniques and exercise program | Change From Baseline at 3 and 6 months in: symptomatology, frequency, and duration of ACTs performance, as well as frequency and duration of exercise program performed
  Compliance with the ACTs will be recorded using a detailed diary that includes weekly symptoms, type, frequency, and duration of ACTs performed. For both groups, compliance will be assessed twice a month, following the completion of this diary. The DHSG will complete the diary through the website, while the CG will complete it in a paper version via a phone call from the physiotherapist. Furthermore, the DHSG's exercise program compliance will be assessed every second online session through a Microsoft Form diary.

SECONDARY OUTCOMES:
Functional Capacity | Change From Baseline in 6MWT distance at 3 and 6 months
  The 6-minute walking test (6MWT) will be used to assess functional capacity. The participants will be asked to walk as far as possible in a 30-m corridor, and standardized encouragement will be given after each minute. The total walking distance (6MWD) will be recorded.
Exercise Capacity (Chester Step test) | Change From Baseline in CST steps at 3 and 6 months
  CST is a multi-staged test that requires participants to step on and off a 20 or 25cm tall step with no handles at a rate set by a metronome beat, which is continuously increasing. Step heights were chosen to be optimal for children according to their age. It consists of 5 levels, each of two minutes duration. The total number of steps and the maximal level achieved will be recorded.
Respiratory muscle strength | Change From Baseline in MIP and MEP scores at 3 and 6 months
  Maximal inspiratory (MIP) and expiratory (MEP) pressure will be measured using a mouth pressure meter (MicroRPM; MicroMedical) to assess respiratory muscle strength. A maximum value of three efforts with a variation of less than 5% will be recorded for both inspiratory and expiratory pressures. There will be a minute rest between the efforts.
Peripheral muscle strength | Change From Baseline in handgrip scores at 3 and 6 months
  Handgrip strength will be assessed using a hand dynamometer (JAMAR, Patterson Medical, IL, USA). Participants will hold the dynamometer at a 90o angle to their elbow. Three separate efforts for the dominant hand grip (DHG) and three for the non-dominant hand grip (NDHG) will be administered, with 30 seconds of rest between efforts. The highest value in kilograms (kg) for each hand will be recorded.
Physical Activity (Physical Activity Questionnaire for Older Children) | Change From Baseline in PAQ-C Score at 3 and 6 months
  The Physical Activity Questionnaire for Older Children (PAQ-C) is a ten-item self-administered questionnaire that intends to measure physical activity (PA). Nine of the ten items are scored on a five-point rating scale, where higher scores indicate a higher level of activity. The first item of the PAQ-C consists of 22 common sports and leisure activities for which the participants select the score based on the frequency of the activities performed during the preceding seven days on a five-point rating scale (1= no activity at all, 2= 1-2 times, 3= 3-4 times, 4= 5-6 times and 5= 7 times or more) after a mean composite score is calculated. The remaining eight items address PA performed during the day (e.g., physical education classes, recess time, lunchtime, as well as after-school activities on weekday evenings and weekends), and a summary for all days of the week. The mean score of the first nine items is the summary score of the PAQ-C.
Physical Activity and Sedentary Behavior (Youth Activity Profile) | Change From Baseline in YAP Score at 3 and 6 months
  The Youth Activity Profile (YAP) comprises 15 items in total, each scored on a 5-point scale designed to capture four components in youth behaviors: 1) PA in school, 2) PA out of school, 3) PA over the weekend, and 4) sedentary behaviors. Each YAP section is developed to be scored independently (ie, items for each dimension score would reflect a higher expected activity levels/sedentary time at that same dimension).
Health-Related Quality of Life | Change From Baseline in PedsQL Score at 3 and 6 months
  Pediatric Quality of Life Inventory Version 4.0 (PedsQL) is a self-administrated questionnaire that includes 23 items divided into four subscales: Physical Functioning (PH), Emotional Functioning (EM), Social Functioning (SOC), and School Functioning (SCH). Responses are given on a five-point scale ranging from 0 (never a problem) to 4 (almost always a problem) and are reverse-scored so that lower scores reflect more negative functioning.
Cough-specific Quality of Life | Change From Baseline in CC-QoL Score at 3 and 6 months
  The Cough-specific Quality of Life (CC-QoL) is a 7-day recall questionnaire designed to reflect several domains related to a child's cough, including physical (e.g., coughing makes you feel tired), social (e.g., others staring at you), and psychological (e.g., feeling upset). The responses are rated on a 7-point Likert scale (1=all the time to 7=none of the time) with higher scores reflecting higher QoL.
Sleep Quality | Change From Baseline in PSQ Score at 3 and 6 months
  The Pediatric Sleep Questionnaire (PSQ) is a tool used to assess sleep-related breathing disorders in children, such as snoring, daytime sleepiness, and related behavioral disturbances. It consists of 22 items with yes/no/don't know responses. Total score consists of the "yes" responses divided by the total number of items (excluding the "don't know" responses).
Digital Health Services Satisfaction | TUQ Score after 12 weeks (end of the intervention)
  Satisfaction from the use of the Vsee platform and FysΑΩ website will be assessed using the Telemedicine Usability Questionnaire (TUQ). The TUQ consists of 21 questions, scored on a Likert scale from 1 (totally disagree) to 7 (totally agree). The total score is calculated by the mean of all 21 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni A Kortianou, Professor, Study Director — Clinical Exercise Physiology and Rehabilitation Research Laboratory; Eleni Kortianou, Professor, Study Chair — Clinical Exercise Physiology and Rehabilitation Research Laboratory; Aspasia Mavronasou, PT, MSc, PhD candidate, Principal Investigator — Clinical Exercise Physiology and Rehabilitation Research Laboratory
Locations (1):
- Physiotherapy Department, University of Thessaly, Lamia, Fthiotis, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180